CLINICAL TRIAL: NCT04602078
Title: Phase II, Multicenter, Non-randomized, Single-arm, Open-label Trial of Atezolizumab in Combination of Split-doses of Gemcitabine Plus Cisplatin in Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Study of Atezolizumab Combined With Split-dose Gemcitabine Plus Cisplatin in Urothelial Carcinoma
Acronym: AUREA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2020-IEC(VEJ)-1; 2020-001326-65 (EudraCT Number)
Record Dates: First submitted 2020-10-06; First posted 2020-10-26 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced or Metastatic Urothelial Carcinoma
Keywords: Cancer; Bladder; Urethra; Ureter; metastatic or locally advanced
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms; Neoplasm Metastasis | interventions — atezolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AUREA single-arm (Experimental): Atezolizumab (1200 mg) intravenously administered every 21 days (one cycle) up to disease progression, unacceptable toxicity or absence of clinical benefit.
  Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle plus Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.
  Interventions: Drug: Atezolizumab 1200 mg/m2; Drug: Gemcitabine 1000 mg/m2; Drug: Cisplatin 70 mg/m2

INTERVENTIONS:
Drug: Atezolizumab 1200 mg/m2 — Fixed dose of 1200 mg/m2 by intravenous (IV) infusion on D1 of each cycle up to disease progression, unacceptable toxicity or absence of clinical benefit.
  Other Names: Tecentriq
Drug: Gemcitabine 1000 mg/m2 — Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle for up to 6 cycles.
Drug: Cisplatin 70 mg/m2 — Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.

SUMMARY:
Phase II, multicenter, non-randomized, single-arm, open-label trial of atezolizumab in combination of split-doses of gemcitabine plus cisplatin in patients with locally advanced or metastatic urothelial carcinoma.

The Aurea trial aims to evaluate the preliminary efficacy of atezolizumab plus split-dose gemcitabine and cisplatin (GC) for the first-line setting, in patients with histologically confirmed advanced (locally advanced and metastatic) urothelial cancer in terms of overall response rate (ORR) assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

Secondary objectives include: efficacy (clinical benefit rate, duration of response, time to response, overall survival and progression-free survival); safety (frequency and severity of adverse events assessed by NCI CTCAE v5.0) and exploratory endpoints ( correlation of prognostic biomarkers/factors with efficacy and relationship between the expression of PD-L1 and microbiome with ORR and PFS).

At least 66 patients will be included.

The treatment schedule is as follows:

Atezolizumab at a fixed dose of 1200 mg/m2 by intravenous (IV) infusion on D1 of each 21-day cycle up to disease progression, unacceptable toxicity or absence of clinical benefit.

Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle plus Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.

DETAILED DESCRIPTION:
The results of trials combining checkpoint inhibitors or platinum-based chemotherapy plus PD-1/PD-L1 inhibitors are eagerly awaited. The combination of split cisplatin with atezolizumab is a feasible treatment that may provide better outcomes than carboplatin/based combinations.

In the IMvigor130, 52% of patients considered cisplatin eligible at the entry of the study were treated with carboplatin. Subanalysis presented at European Society of Medical Oncology (ESMO) 2019 (Grande E, et al. 2019) has also shown a longer median OS are achieved with cisplatin-based chemotherapy combined with atezolizumab (21.7 months) when compared to the carboplatin-based chemotherapy plus atezolizumab (14.2 months), with similar findings when it comes to PFS 8.8 months with cisplatin/gemcitabine/atezolizumab vs 7.1 months carboplatin/gemcitabine/atezolizumab.

A reasonable strategy may be the use of split cisplatin with atezolizumab to increase the number of patients receiving cisplatin.

The AUREA study is a multicenter, open labelled, single arm, multicohort Phase II clinical trial of of atezolizumab in combination of split-dose cisplatin plus gemcitabine in patients with locally advanced or metastatic urothelial carcinoma (additional details on the eligibility criteria of the study are found in section 6 of this protocol).

The design includes screening phase, combined treatment initial phase, monotherapy treatment phase, follow-up phase and translational research with biopsies, blood samples and faecal samples.

The dose scheme includes the initial dose of atezolizumab (1200 mg) intravenously administered every 21 days (one cycle) up to disease progression, unacceptable toxicity or absence of clinical benefit. Dose adjustment or dose reductions of atezolizumab are not expected. AUREA is an Investigator Initiated Study, the Sponsor will supply Atezolizumab for up to 24 months of treatment for each patient. For those patients in which the PI considers that the best option for the patient is continuing atezolizumab for more than 24 months, available commercial Site supplies should be used, after managed local administrative regulation. Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle plus Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.

Study treatment will begin as soon as possible after signing the informed consent. Before each treatment administration chemotherapy/atezolizumab administration laboratory, medical consulting and other determinations will be performed to ensure that treatment can be safely administered.

A CT Scan or MRI will be performed at baseline, on week 9, week 18 and then every 12 weeks (q12w) ± 1w until objective disease progression as per PI's criteria or death (whichever comes first). Blood samples for biomarkers studies should be collected before administration of cycle 4 and at the time of Progression Disease (PD) (end of treatment if applicable).

For patients with progression reported as per RECIST criteria at week 9, continuity of treatment with atezolizumab should be evaluated by the PI of each site as per clinical benefit criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 18 years old.
2. Written informed consent approved by the Independent Ethics Committee (IEC), prior to the performance of any trial activities.
3. Patients with histologically documented, locally advanced (T4B, any N; or any T, N2-3) or metastatic urothelial carcinoma (M1, Stage IV)*.

   *Also termed transitional cell carcinoma (TCC) or Urothelial Cell Carcinoma (UCC) of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra).
4. Patients should not be eligible (unfit) for full dose of cisplatin, in the investigator's judgement, based on:

   a. Age older than 70 years. b. Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 2 or Karnofsky PS of 60 - 70% (only 15 patients will be included with ECOG 2). c. Measured creatinine clearance (ClCr) > 30 and < 60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for the determination of creatinine clearance:

   Males:

   Creatinine Clearance (CL) (mL/min) = Weight (kg) × (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) =

   Weight (kg) × (140 - Age) ×0.85 72 x serum creatinine (mg/dL) d. Any other reason the physician considers but should specify in the Case Report Form (CRF) and discussed with the PI.
5. At least one measurable lesion through radiographic tumor evaluation (CT scan or magnetic resonance imaging/MRI) as defined by RECIST version 1.1, that has not been previously irradiated within 4 weeks prior to the study enrolment.
6. Patients with an archival or de novo tumor biopsy (representative formalin-fixed paraffin-embedded (FFPE) paraffin block obtained within 6 months prior to inclusion) with an associated pathology report, for testing of PD-L1 expression prior to study enrollment. Samples in unstained slides could be acceptable (at least 15 slides).
7. Patients with adequate normal organ and marrow function as defined below:

   1. Haemoglobin ≥ 9.0 g/dL.
   2. Absolute neutrophil count (ANC) > 1500 per mm
   3. Platelet count ≥ 100,000 per mm
   4. Serum bilirubin ≤ 1.5 X institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be ≤ 2X ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of haemolysis or hepatic pathology); however, they will be allowed only in consultation with their physician.
   5. Serum transaminases (ALT, AST and GGT) ≤ 2.5X institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 3X ULN.
8. No major active bleeding.
9. Female subjects of childbearing potential (not surgically sterile or at least 2 years postmenopausal) must provide a negative urine pregnancy test at screening, and use a medically accepted double barrier method of contraception. In addition, they must agree to continue the use of this double barrier method for the duration of the study and for 6 months after participation in the study.
10. Males should agree to abstain from sexual intercourse with a female partner or agree to use a double barrier method of contraception (i.e. condom with spermicide, in addition to having their female partner use some contraceptive measures such as oral contraceptive drugs, intrauterine device (IUD) hormonal contraception, or cervical caps), for the duration of the study and for 6 months after participation in the study
11. Willingness and ability of patients to comply with the protocol for the duration of the study including undergoing treatment as well as availability for scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Prior treatment with any immune checkpoint inhibitor therapy (e.g., CTLA4, PD-1, or PD-L1 targeting agent).*
2. Presence of active second malignancy and/or prior malignancy in the last 2 years is allowed except for the following:

   1. adequately treated basal cell or squamous cell skin cancer,
   2. adequately treated Stage I or II cancer from which the patient is currently in complete remission per investigators' clinical judgment.
3. Patient receiving radiation therapy within 4 weeks before inclusion.
4. Active or prior documented autoimmune disease within the past 2 years. Note:

   Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
5. Active or prior documented inflammatory bowel disease (e.g.., Crohn's disease and ulcerative colitis).
6. History of allogeneic organ transplant.
7. Subjects having a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment.
8. Current or prior use of immunosuppressive medication within 7 days prior to enrolment, except the following:

   a. Intranasal, inhaled, topical steroids, or local steroid injections i. Systemic corticosteroids at physiologic doses ≤10 mg/day of prednisone or equivalent; ii. Steroids as premedication for hypersensitivity reactions
9. The subject has uncontrolled, significant intercurrent or recent illness (within 6 months prior to inclusion) including, but not limited to, the following conditions:

   a. Cardiovascular disorders: i. Class 3 or 4 congestive heart failure as defined by the New York Heart Association, unstable angina pectoris, and serious cardiac arrhythmias. ii. Uncontrolled hypertension defined as sustained blood press > 150 mm hg systolic or > 100 mm hg diastolic despite optimal antihypertensive treatment. iii. Stroke (including Transient Ischemic Attack (TIA)), myocardial infarction, other ischemic event, or thromboembolic event within 6 months before inclusion. Subjects with a more recent diagnosis of Deep Vein Thrombosis (DVT) are allowed if stable, asymptomatic, and treated with Low Molecular Weight Heparin (LMWH) for at least 6 weeks before study treatment.

   b. Gastrointestinal disorders (e.g., malabsorption syndrome or gastric outlet obstruction) including those associated with a high risk of perforation or fistula formulation: i. Tumours invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction. ii. Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before inclusion. Note: complete healing of an intra-abdominal abscess must be confirmed prior to start of the treatment.

   c. Clinically significant hematemesis or hemoptysis of > 0.5 teaspoon (> 2.5 ml) of red blood or history of other significant bleeding within 3 months before treatment.

   d. Cavitating pulmonary lesion(s) or known endobronchial disease manifestation.

   e. Lesions invading major pulmonary blood vessels.

   f. Other clinically significant disorders such as: i. Active infection requiring systemic treatment, infection with human immunodeficiency virus or acquired immunodeficiency syndrome-related illness, or chronic hepatitis B or C infection.

   ii. Serious non-healing wound/ulcer/bone fracture. iii. Malabsorption syndrome. iv. Moderate to severe hepatic impairment (child-pugh B or C). v. Requirement for hemodialysis or peritoneal dialysis. vi. Uncontrolled diabetes mellitus.
10. Major surgery (e.g., GI surgery and removal or biopsy of brain metastasis) within 8 weeks before inclusion. Complete wound healing from major surgery must have occurred 4 weeks before study treatment and from minor surgery at least 10 days before study treatment. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
11. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
12. Any test for hepatitis B virus (HBV) or hepatitis C virus (HCV) indicating acute or chronic infection.
13. Women who are pregnant or are breastfeeding.
14. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy.
15. Any of the following within 6 months prior to study entry: myocardial infarction, uncontrolled angina, uncontrolled hypertension, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
16. Previously identified allergy or hypersensitivity to components of the study treatment formulations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Velasco, M.D., Ph.D., Study Chair — Hospital Universitario 12 de Octubre
Locations (12):
- Spain (12):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO Hospitalet- Hospital Duran i Reynals, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario de Jaén, Jaén
  - Complejo Hospitalario Universitario Insular Marterno Infantil, Las Palmas de Gran Canaria
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Universitario Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Virgen de la Salud, Toledo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients screened
Groups:
- AUREA Single-arm: Atezolizumab (1200 mg) intravenously administered every 21 days (one cycle) up to disease progression, unacceptable toxicity or absence of clinical benefit.
  Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle plus Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.
  Atezolizumab 1200 mg/m2: Fixed dose of 1200 mg/m2 by intravenous (IV) infusion on D1 of each cycle up to disease progression, unacceptable toxicity or absence of clinical benefit.
  Gemcitabine 1000 mg/m2: Gemcitabine 1000 mg/m2 IV on D1 and 1000 mg/m2 IV on D8 of each 21-day cycle for up to 6 cycles.
  Cisplatin 70 mg/m2: Cisplatin 70 mg/m2 by IV on split-dose schedule of 35 mg/m2 on day 1 (D1) and 35 mg/m2 on day 8 (D8) for up to 6 cycles.
Period: Overall Study
Arm/Group | AUREA Single-arm
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 71 [49 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 57
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 66
Eastern Cooperative Oncology Group performance status (ECOG-PS) [Count of Participants; unit: Participants] — Scale validated by the World Health Organization (WHO) to assess the quality of life of cancer patients. The scale ranges from 0, patient fully active, to 5, patient dead.
  Participants
    Score 0 | 17
    Score 1 | 34
    Score 2 | 15
Site of the primary tumor [Count of Participants; unit: Participants] — Location of the primary tumor in the genitourinary tract: The upper tract was defined as the renal pelvis or ureter, and the lower tract as the bladder and urethra.
  Participants
    Upper tract | 11
    Lower tract | 55
Stage at inclusion [Count of Participants; unit: Participants] — Measures the extend of spread of the disease at the time of inclusion
  Participants
    Locally advanced | 8
    Metastatic | 58
Metastatic locations [Count of Participants; unit: Participants] — Percentage of patients with organs affected by the disease. A patient may have more than 1 oragan affected
  Participants
    Lymph nodes: Affected | 44
    Lymph nodes: Not affected | 22
    Lung: Affected | 36
    Lung: Not affected | 30
    Bone: Affected | 20
    Bone: Not affected | 46
    Liver: Affected | 12
    Liver: Not affected | 54
Reason unfit for full dose chemotherapy [Count of Participants; unit: Participants] — Criteria to consider patients not eligible for full doses of cisplatin. A patient may have more than one reason to be considered ineligible.
  Participants
    ECOG 2: Yes | 15
    ECOG 2: No | 51
    Age > 70 years: Yes | 36
    Age > 70 years: No | 30
    creatinine clearance 30-60 μmol/L: Yes | 33
    creatinine clearance 30-60 μmol/L: No | 33
Prior local therapy [Count of Participants; unit: Participants]
  Surgery: Yes | 58
  Surgery: No | 8
  Radiotherapy: Yes | 9
  Radiotherapy: No | 57
PD-L1 status [Count of Participants; unit: Participants] — PD-L1, quantified using immunohistochemistry assays, is currently the most widely validated, used and accepted biomarker to guide the selection of patients to receive immunotherapy such as atezolizumab in this trial.
  Positivity indicates high expression of this biomarker and it has been shown to correlate with eficacy of immunotherapy in some tumor types. Negativity usually correlatess with worse prognosis to immunotherapy.
  The prognostic value of PL-L1 in many cancer types is still under study.
  Participants
    Positive | 14
    Negative | 26
    Unknown | 26

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period according to RECIST 1.1 criteria. Evaluated by Computed tomography scans (CT scan).
Time Frame: Through study completion, average 2 years.
Measure: Number (95% Confidence Interval); unit: Percentage of patients with response
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Percentage of patients with response | 48.5 [36 to 61.1]

2. Secondary Outcome: Duration of Response (DoR)
Description: Time from first confirmed response (CR or PR) to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first.
Time Frame: Through study completion, average 2 years. CT scans for evaluation will be performed at baseline, on week 9, week 18 and then every 12 weeks (q12w) ± 1w until objective disease progression
Population: Patients with CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 32
months | 9.2 [5.5 to 16.8]

3. Secondary Outcome: Time to Response (TtR)
Description: Time from first dosing date to the date of the documented ORR as determined using RECIST 1.1 criteria.
Time Frame: Through study completion, average 2 years. CT scans for evaluation will be performed at baseline, on week 9, week 18 and then every 12 weeks (q12w) ± 1w until objective disease progression as per PI's criteria or death (whichever comes first).
Population: Patients with CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 32
months | 2.1 [2 to 2.2]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Percentage/proportion of patients with confirmed complete response (CR) or partial response (PR), or stable disease (SD) as their overall best response throughout the study period.
Time Frame: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of patients with response
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Percentage of patients with response | 66.7 [54 to 77.8]

5. Secondary Outcome: Overall Survival (OS)
Description: Time from first dosing date to the date of death. A subject who has not died will be censored at the last known date alive.
Time Frame: Through study completion, average 2 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
months | 12.9 [10.2 to 20.2]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from first dosing date to the date of confirmed PD. A subject who has not died will be censored at the last known date alive.
Time Frame: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
months | 6.9 [6.7 to 9.4]

7. Secondary Outcome: 6 Months Progression-Free Survival (PFS)
Description: Proportion of patients free of PD at 6 months since start of treatment. A subject who has not died will be censored at the last known date alive.
Time Frame: 6 months from the first dose administration. CT scans for evaluation will be performed at baseline, on week 9, week 18 and then every 12 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Percentage of patients | 67.6 [57.1 to 80]

8. Secondary Outcome: Adverse Events Frequency (Safety)
Description: Frequency of adverse events (AEs) reported classified by type and severity.
Time Frame: Through study completion, average 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Participants
  Any grade AE: Experienced AEs | 66
  Any grade AE: Did not experience AEs | 0
  AE Grade >=3: Experienced AEs | 62
  AE Grade >=3: Did not experience AEs | 4

9. Secondary Outcome: Treatment-related Adverse Events Frequency (Safety)
Description: Frequency of treatment-related adverse events reported classified by type and severity.
Time Frame: Through study completion, average 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 66
Participants
  Treatment-related AEs any grade: Experienced AEs | 62
  Treatment-related AEs any grade: Did not experience AEs | 4
  Treatment-related AEs grade >=3: Experienced AEs | 44
  Treatment-related AEs grade >=3: Did not experience AEs | 22

10. Other Pre Specified Outcome: Progression Free Survival Measured by RECIST 1.1 in Patients Grouped According to Their PD-L1 Expression
Description: Correlation between the expression of PD-L1 with PFS during experimental treatment. Patients will be grouped based on the PD-L1 expression levels in PD-L1 positive or negative patients. Progression free survival will be assessed in both groups of patients and compared to identify potential statistically significant differences between groups.
Time Frame: PD-L1 expression measured at the end of the trial. PFS assessed Through study completion, average 2 years
Population: 26 patients had no PD-L1 determined
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 40
months
  PD-L1 positive: number analyzed (Participants) | 14
  PD-L1 positive | 6.9 [6.4 to 17]
  PD-L1 negative: number analyzed (Participants) | 26
  PD-L1 negative | 6.9 [6 to 9.7]
Statistical Analysis 1: Comparison: AUREA Single-arm; Comparisong between subgroups: patients with PD-L1 postive versus patients with PD-L1 negative; Test type: Superiority; p = 0.444, Log Rank

11. Other Pre Specified Outcome: ORR Measured by RECIST 1.1. in Patients Grouped According to Their PD-L1 Expression
Description: Correlation between the expression of PD-L1 with ORR during experimental treatment. Patients will be grouped based on the PD-L1 expression levels in PD-L1 positive or negative patients. ORR will be assessed in both groups of patients and compared to identify potential statistically significant differences between groups.
Time Frame: PD-L1 expression measured at the end of the trial. ORR assessed Through study completion, average 2 years
Population: 26 patients had no PD-L1 determined
Measure: Count of Participants; unit: Participants
Arm/Group | AUREA Single-arm
Number analyzed (Participants) | 40
Participants
  PD-L1 positive: number analyzed (Participants) | 14
  PD-L1 positive: Tumor objective response | 8
  PD-L1 positive: No response | 6
  PD-L1 negative: number analyzed (Participants) | 26
  PD-L1 negative: Tumor objective response | 10
  PD-L1 negative: No response | 16
Statistical Analysis 1: Comparison: AUREA Single-arm; Comparisong between subgroups: patients with PD-L1 postive versus patients with PD-L1 negative; Test type: Superiority; p = 0.414, Chi-squared

ADVERSE EVENTS:
Time Frame: Through study completion, average 2 years.
Arm/Group | AUREA Single-arm
All-Cause Mortality (participants affected / at risk) | 47/66
Serious Adverse Events (participants affected / at risk) | 48/66
Other Adverse Events (participants affected / at risk) | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUREA Single-arm (N=66)
Abdominal pain (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (6)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Pancitopenia (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Death NOS (General disorders) | 1 (1)
Disease progression (General disorders) | 18 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Incarcerated hernia (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 3 (5)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
traumatic head injury (Injury, poisoning and procedural complications) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Inmune-mediated myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Traumatic brain injury (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (2)
Acute nephritis (Renal and urinary disorders) | 1 (2)
Nephritis (Renal and urinary disorders) | 1 (1)
Acute pyelonephritis (Renal and urinary disorders) | 1 (1)
Impaired renal function (Renal and urinary disorders) | 1 (1)
COVID 19 (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
left percutaneous nephrostomy non-permeable (Surgical and medical procedures) | 1 (1)
Bladder TUR (Surgical and medical procedures) | 1 (1)
Urethral TUR (Surgical and medical procedures) | 1 (1)
Prostate TUR (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 10 (12)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Bilateral Pulmonary Embolism (Vascular disorders) | 1 (1)
Hemorragic hipovolemic shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AUREA Single-arm (N=66)
Abdominal pain (Gastrointestinal disorders) | 6
Anemia (Blood and lymphatic system disorders) | 43
Anorexia (Metabolism and nutrition disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (General disorders) | 9
Constipation (Gastrointestinal disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 7
Diarrhea (Gastrointestinal disorders) | 10
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 4
Edema limbs (Respiratory, thoracic and mediastinal disorders) | 6
Fatigue (General disorders) | 41
Fever (General disorders) | 9
Hematuria (Renal and urinary disorders) | 13
Hyperglycemia (Investigations) | 6
Hypomagnesemia (Investigations) | 8
Hypothyroidism (Endocrine disorders) | 9
Insomnia (Psychiatric disorders) | 6
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 24
Neutrophil count decreased (Blood and lymphatic system disorders) | 33
Pain in extremity (General disorders) | 10
Platelet count decreased (Blood and lymphatic system disorders) | 26
Pruritus (Skin and subcutaneous tissue disorders) | 6
COVID-19 (Infections and infestations) | 6
Serum amylase increased (Investigations) | 6
Tinnitus (Ear and labyrinth disorders) | 7
Urinary tract infection (Renal and urinary disorders) | 17
Vomiting (Gastrointestinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT04602078/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT04602078/SAP_001.pdf